CLINICAL TRIAL: NCT04546880
Title: Effects of Breathing Exercises in the Mothers of Children With Special Health Care Needs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hasan Kalyoncu University (Other)
Responsible Party: Principal Investigator, Aysenur Tuncer, Assistant Professor, Hasan Kalyoncu University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HKUatuncer
Record Dates: First submitted 2020-08-29; First posted 2020-09-14 (Actual); Last update posted 2020-09-14 (Actual); Status verified 2020-09

CONDITIONS: Chronic Low-back Pain
Keywords: Chronic Low back pain; Breathing exercises; Core Stabilization; Anxiety; Sleep
MeSH Terms: conditions — Anxiety Disorders | interventions — Breathing Exercises

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1:Breathing and Stabilization Exercise Group (Experimental): Breathing exercises combined with stabilization exercises
  Interventions: Other: Breathing exercises; Other: Stabilization exercises
- Group 2: Stabilization Exercise Group (Active Comparator): Only Stabilization exercises therapy
  Interventions: Other: Stabilization exercises

INTERVENTIONS:
Other: Breathing exercises — Breathing exercises consist of the techniques of diaphragmatic and pursed-lip breathing. During the diaphragmatic breathing, attention is focused on the correct abdominal breathing.
  The pursed-lip breathing is one step further to the diaphragmatic breathing and a technique designed to have control time and volume over breathing.
  Arms: Group 1:Breathing and Stabilization Exercise Group
Other: Stabilization exercises — Training about the concepts of stabilization and abdominal bracing is given before starting to the study. The motor control tests for local muscles transversus abdominus and multifidi are performed after the training. The abdominal bracing test is performed in the quadruped position, in prone, and in hook lying position with the patient's spine supine with hips and knees flexed and knees in contact with the surface.
  The second stage consists of closed-chain segmental control exercises. It is a series of weight-bearing exercises are performed on stable and unstable surfaces. The last stage of the stabilization program is an open kinetic chain exercise to promote distal stability.

SUMMARY:
The aim of the study is to determine the effectiveness of breathing exercises combined with core stabilization exercises in mothers with chronic non-specific low back pain of children with special health care needs.

DETAILED DESCRIPTION:
A total of 46 mothers having children with special health care needs participate in the study.

Twenty-three mothers in the experimental group receive stabilization exercises with breathing exercises 3 times a week for 8 weeks while 23 mothers in the control group receive only stabilization exercises during the same period of time. Each exercise session lasts about 60 minutes and was performed 3 days per week, for 8 weeks. All mothers in both groups perform 15 minutes warm-up stretching exercises prior to the core exercises and 10 minutes cool-down exercises at the end of each session.

Breathing with the stabilization exercise group receives breathing exercises before the stabilization exercise program. A one-hour theoretical training is given to the mothers about the techniques of diaphragmatic and pursed-lip breathing at the beginning of the study. The pursed-lip breathing is one step further to the diaphragmatic breathing. Patients are instructed to do breathing exercises during the stabilization exercises, in which patients focus on their breathing circle, time, and movement while doing the stabilization exercises.

All 46 mothers in both groups are given a one-hour training about the stabilization exercises before starting the study. The motor control tests for local muscles transversus abdominus and multifidi are performed after the training. The abdominal bracing test is performed in the quadruped position, in prone, and in hook lying position with the patient's spine supine with hips and knees flexed and knees in contact with the surface. Closed-chain segmental control exercises, a series of weight-bearing exercises, and open kinetic chain exercises to promote distal stability are performed.

ELIGIBILITY:
Inclusion Criteria:

* Primary caregiver of the child
* Suffering from LBP for at least three months
* Lumbar instability
* Absence of radiculopathy or other damages to the spine
* Not receiving any types of physical therapy during the trial or at least six months prior to the study
* Enough physical autonomy to participate in the physical activities
* Be volunteer
* Be compliant for the study

Exclusion Criteria:

* Taking any anti-depressant medications and/or having psychotherapy
* Any surgery within the last 3 months
* Be pregnant
* Presence of dysfunction of the musculoskeletal system during the study
* Participation rate lower than 80% of the program schedule

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 46 (Actual)
Dates: Start 2018-06-15 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2019-02-20 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Low Back Pain at 8 weeks | Baseline, 8 weeks
  Visual Analog Scale were used where patients were asked to rate their pain on a scale from 0 to 10 with 0 indicating no pain and 10 the maximum worst pain at the baseline and the end of 8 weeks intervention.
Change from Baseline in Fatigue at 8 weeks | Baseline, 8 weeks
  Fatigue Severity Scale was used where patients were asked to indicate their levels of agreement with a 0-7 scale indicating "0" strong disagreement and "7" strong agreement at a total of 9 questions. A sum of all responses was calculated for analysis. Sixty-three was the maximum score. The higher value represented a higher level of fatigue.
Change from Baseline in Anxiety at 8 weeks | Baseline, 8 weeks
  Spielberger's State-Trait Anxiety Inventory was used to measure state and trait anxiety with 20 item self-report rating scale. The range of total scores was 20-80, and higher scores indicated higher levels of anxiety.
Change from Baseline in Sleep quality at 8 weeks | Baseline, 8 weeks
  Pittsburg Sleep Quality Index was used to assess sleep quality consisting of a total of 24 questions, 19 of which were self-rated by the patient, and 5 of which were answered by the partner of the patient. The total scores ranged between 0 and 21 points with higher values representing worse sleep quality.

CONTACTS AND LOCATIONS:
Locations (1):
- Hasan Kalyoncu University, Gaziantep, Turkey (Türkiye)